CLINICAL TRIAL: NCT04472910
Title: GATA6 Expression as a Predictor of Response to Peri-Operative Chemotherapy in Resectable Pancreatic Adenocarcinoma: A Multicentre Canadian Phase II Study
Brief Title: GATA6 Expression as a Predictor of Response to Peri-Operative Chemotherapy in Resectable Pancreatic Adenocarcinoma
Acronym: NeoPancOne
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Pancreatic Cancer Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-6059
Record Dates: First submitted 2020-06-23; First posted 2020-07-16 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Resectable Pancreatic Cancer
MeSH Terms: interventions — folfirinox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Neo-adjuvant mFFX (Experimental): Neo-adjuvant mFFX up to 6 cycles, surgery, adjuvant chemotherapy for up tp 6 cycles, follow up
  Interventions: Drug: Modified Folforinox (mFFX)

INTERVENTIONS:
Drug: Modified Folforinox (mFFX) — Neo-adjuvant mFFX for up to 6 cycles, chemo-Adjuvant FFX q 2 weekly or other approach as per investigator to complete up to 6 months chemotherapy
  Other Names: Folfirinox or other approach

SUMMARY:
To date, there have been no Canadian led neoadjuvant or peri-operative trials, this multicentre design gives the opportunity to build more experience with this strategy across Canada in more institutions. The design of this prospective trial will also test our important hypotheses regarding the use of biomarkers to understand the benefit of mFFX in improving outcomes for patients with resectable pancreas cancer. Data from this study would likely inform future studies where patients are given personalised options for the best treatment strategies rather than one empiric approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological diagnosis of PDAC. Those with unconfirmed histology must have this confirmed by EUS-FNB in the pre-screening period prior to commencement of chemotherapy. Invasive PDAC in the setting of intraductal papillary mucinous neoplasm (IPMN) is permitted.
* Patients must consent to EUS-FNB for correlative analysis even if adenocarcinoma has been confirmed, unless confirmation was performed using a previous biopsy or fine needle biopsy with adequate tumour tissue for GATA6 analysis.
* Resectable primary tumour on preoperative biphasic (arterial and venous phases) contrast-enhanced CT for pancreatic staging as per institutional standard of care, with ≤5 mm slice thickness. MRI for liver metastases (optional) as per institutional standard of care. The definition of resectability (as per NCCN guidelines - see Appendix B) includes:

  * no involvement of the celiac artery, common hepatic artery or superior mesenteric artery (or if present a replaced right or common hepatic artery)
  * no involvement or <180 (interface between tumour and vessel wall, of the portal vein or superior mesenteric vein, and patent portal vein/splenic vein confluence_
  * For tumours of the body and tail of the pancreas, involvement of the splenic artery and vein of any degree is considered resectable disease
* Patients must be medically fit to undergo surgical resection
* No prior oncological treatment for index PDAC
* ECOG Performance status 0-1
* Age > 18 years
* Patients must be medically suitable for treatment with mFFX as per treating medical oncologist
* No evidence of metastases (i.e., metastatic work-up negative including a CT scan of the chest, abdomen (IV and oral contrast, 3 phase) and pelvis)
* Adequate hematologic function

  * absolute neutrophil count (ANC) ≥ 1,500 cells/mm3
  * platelets ≥ 100 000 cells/mm3
  * hemoglobin ≥ 9 g/L (after transfusion is acceptable))
* Creatinine level < 130 µmol/L or CrCl ≥ 50 ml/min
* Patients of child-bearing potential (for female patient: study entry after a menstrual period and a negative pregnancy test) must agree to use two medically acceptable methods of contraception (one for the patient and one for their partner) during the study and for 4 months after the last study treatment intake for women and 6 months for men. These patients must have a pregnancy test repeated every month while on chemotherapy.
* Patients must be able to provide written informed consent
* Adequate liver function (AST <2.5 times the institutional upper limit of normal at the baseline visit, total bilirubin ≤ 2 times the institutional upper limit of normal at the baseline visit)

Exclusion Criteria:

* Patients where attempted EUS-FNB x 2 has not confirmed PDAC in the setting of unconfirmed histology.
* Patients in whom histology has confirmed PDAC but who do not consent to EUS-FNB, unless previous confirmation was by biopsy or fine needle biopsy with adequate tumour tissue for GATA6 analysis.
* Non-ductal pancreas tumours including endocrine tumours, acinar cell carcinoma, cyst adenocarcinoma or ampullary tumours.
* Unresectable PDAC by contrast enhanced CT or MRI. Borderline resectable PDAC (vein and artery) are excluded from this study
* Evidence of metastatic disease
* Prior treatment for index PDAC
* Previous autologous bone marrow transplant or stem cell rescue
* Active hepatitis B or C infection
* Uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* History of another primary cancer within the last 3 years with the exception of non-melanoma skin cancer, early stage prostate cancer or curatively treated cervical carcinoma in situ or other indolent malignancy (discretion of PI).
* Pregnant or breast-feeding patients are excluded from this study as the chemotherapy agents used in this study have been demonstrated or have the potential to be teratogenic and there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother
* Patients who are being therapeutically anticoagulated with coumadin and cannot have an alternative anticoagulation regimen.
* Known hypersensitivity to any of the drugs used or their components.
* Patients with known complete absence of dihydropyrimidine dehydrogenase (DPD) activity.
* History of QT prolongation or receiving QT prolonging medications.
* History of Gilberts condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-08-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess disease free survival (DFS) in resectable PDAC treated with peri-operative mFFX according to baseline GATA6 expression level | 2-4 years
  Disease free survival

SECONDARY OUTCOMES:
Evaluate the feasibility of EUS FNB as an effective modality for the detection of GATA6 expression at first diagnosis, including number of unsuccessful EUS-FNBs. | 2-4 years
Determine GATA6 in-situ hybridization (ISH)/immunohistochemistry (IHC) success rate | 2-4 years
Determine GATA6 expression levels in EUS-FNB specimen compared to surgical specimen | 2-4 years
Determine the DFS according to R0 or R1 resection status | 2-4 years
Determine the DFS according to baseline Ca19.9 levels | 2-4 years
Determine the DFS according to modified Moffitt RNA classification | 2-4 years
To determine the overall response rate (ORR) to neoadjuvant mFFX | 2-4 years
Determine the percentage of patients who progress on neoadjuvant mFFX | 2-4 years
Assess pathological response rate to mFFX in the neoadjuvant setting | 2-4 years
Determine the overall survival (OS) according to GATA6 expression level in the overall population and the GATA6 high/low populations | 2-4 years
Determine the overall survival (OS) according to R0/R1 resection status in the overall population and the GATA6 high/low populations | 2-4 years
Determine the overall survival (OS) according to baseline Ca19.9 levels in the overall population and the GATA6 high/low populations | 2-4 years
Determine the overall survival (OS) according modified Moffitt classification in the overall population and the GATA6 high/low populations | 2-4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, MD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (8):
- Canada (8):
  - BC Cancer Agency Vancouver, Vancouver, British Columbia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Sunnybrook Hospital/Odette Cancer Centre, Toronto, Ontario
  - Unity Health (St. Joseph's and St. Michael's), Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No